CLINICAL TRIAL: NCT02018471
Title: Management of Anxiety Related to Diagnostic Screenings: an Exploratory Pilot Study
Brief Title: Psychological Counselling in Diagnostic Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Principal Investigator, Malihe Shams, Psychologist, Istituto Oncologico Veneto IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IOV-2012 ANXIETY
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Cancer
Keywords: anxiety; psychoeducational training; coping; relaxation
MeSH Terms: conditions — Neoplasms; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pilot group (Experimental): Forty-three patients who had to undergo one or more diagnostic tests (PET, TAC, fMRI, Mammography, Endoscopy, Colonoscopy) took part in the study. Most of the 43 patients had to undergo only one diagnostic test, and only 6 patients had more than one. They have attended a psychoeducative training.
  Interventions: Behavioral: Psychoeducative training

INTERVENTIONS:
Behavioral: Psychoeducative training — The Psychological education was inspired by the technique, Systematic Desensitization (SD), a therapeutic procedure that seeks to eliminate fear and avoidance behaviour
  Other Names: Systematic Desensitization; Psychological counseling

SUMMARY:
Diagnostic tests have a deep emotional impact on oncology patients. Anxiety and worries can lead people to avoid screening tests, with high risks for health. A single arm, pilot study was organized to evaluate the feasibility and efficacy of psychological counselling for cancer patients who demonstrated anxiety for diagnostic tests. The hypothesis was that taking part in Psychoeducative Training could offer a new modality to reduce anxiety, before and during tests, and also the possibility to reinforce coping strategies.

DETAILED DESCRIPTION:
The Psychoeducative Training was organized in 6 weekly meetings lasting two hours. Each group was composed of 6 participants. The Training follows the cognitive-behavioural model. In the first part of every meeting, theoretical aspects about stress and anxiety were explained, while in the second part some relaxation techniques were taught. During relaxation, we used a selected music that was also going to be used during the diagnostic tests. Since the first meeting, patients experienced these relaxing techniques in order to learn them. In order to support the adaptability, at the end of every meeting the participants received some homework. They had to take notes on how many times they repeated the relaxation exercises and on the anxiety level before and after the training.

For the study, 43 people were recruited. Anxiety was measured with Beck Anxiety Inventory (BAI); it values the seriousness of the physiological behaviour connected with anxiety. This test an "anxiety gauge", which allows us to obtain numerical data on emotional changes. The test is composed of 4 interpretative levels: serious, moderate, small and minimal anxiety.

The coping style was measured with Coping Orientation to Problems Experienced-New Italian Version (COPE-NIV); this test evaluates the way in which people resolve and face traumatic or usual stressful situations.

The research project was approved by the Ethics Committee of Veneto Institute of Oncology.

Every patient signed a written informed consent to process the data for research purposes and to publish it.

Forty-three patients who had to undergo one or more diagnostic tests (PET, TAC, fMRI, Mammography, Endoscopy, Colonoscopy) took part in the study. The average age was 52.4 and 61.5% were married.

ELIGIBILITY:
Inclusion Criteria:

* age: 25 to 65 years cancer patients who must undergo diagnostic tests: TAC, PET, fMRI, Mammography, Endoscopy and Colonoscopy.
* an anxiety level greater than 5 (in a scale from 0=very calm to 10=very anxious; using a self-reporting instrument created ad hoc)
* signed informed consent

Exclusion Criteria:

* healthy people

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients considered drop-outs | 6 weeks after recruitment (end of treatment)
  The proportion of patients considered drop-outs. A patient is considered a drop-out if he/she does not attend at least 2 out of 6 programmed meetings. This is a feasibility outcome

SECONDARY OUTCOMES:
median BAI score after intervention | 6 weeks after recruitment (end of treatment)
  This is an efficacy outcome
median COPE score - Social support score after intervention | 6 weeks after recruitment (end of treatment)
  This is an efficacy outcome
median COPE score - Avoidance strategies score after intervention | 6 weeks after recruitment (end of treatment)
  This is an efficacy outcome
median COPE score - Positive attitude score after intervention | 6 weeks after recruitment (end of treatment)
  This is an efficacy outcome
median COPE score - Problem acceptance score after intervention | 6 weeks after recruitment (end of treatment)
  This is an efficacy outcome
recruitment time (process) | 6 weeks after recruitment (end of treatment)
  This is a feasibility outcome
mean number of recruited patients per week (process) | 6 weeks after recruitment (end of treatment)
  This is a feasibility outcome
refusal rate among eligible patients (process) | 6 weeks after recruitment (end of treatment)
  This is a feasibility outcome
rate of patients who obviously meet and do not meet the eligibility requirements (process) | 6 weeks after recruitment (end of treatment)
  This is a feasibility outcome
number of questionnaires correctly filled out (process) | 6 weeks after recruitment (end of treatment)
  This is a feasibility outcome
phone lines overloaded or waiting room overcrowded by study participants (management) | 6 weeks after recruitment (end of treatment)
  This is a feasibility outcome

CONTACTS AND LOCATIONS:
Overall Officials: Malihe Shams, Principal Investigator — Istituto Oncologico Veneto IRCCS